CLINICAL TRIAL: NCT01875952
Title: Integral Research of the Managing and Treatment of the Infection With Human Immunodeficiency (VIH) /Human Immunodeficiency Syndrome(SIDA) Co-infection With Latent Tuberculosis Infection. A Multidisciplinary and Interinstitucional Approach
Brief Title: Diagnosis and Treatment of Co-infection With Human Immunodeficiency Virus /Latent Tuberculosis Infection (HIV/TBL)
Acronym: HIV/TB
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: Instituto Nacional de Enfermedades Respiratorias (Other Government); Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Ma. de Lourdes Garcia Garcia, Director of the Center of Research in Infectious Diseases, Instituto Nacional de Salud Publica, Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Informed Consent:552 / 306; 000000000014520 (Other: National Council for Science and Technology (CONACYT))
Record Dates: First submitted 2012-03-28; First posted 2013-06-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Human Immunodeficiency Virus (HIV); Tuberculosis (TB); Latent Tuberculosis Infection (LTI)
Keywords: Latent tuberculosis infection; Human immunodeficiency virus (HIV); Treatment; Isoniazid
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis; Latent Tuberculosis | interventions — Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- one arm (Other): All patients with response to positive purified protein derivative (PPD) test are treated
  Interventions: Drug: Isoniazid

INTERVENTIONS:
Drug: Isoniazid — Isoniazid, 10 mg/Kg/day, no more than 300 mg/day, for six months

SUMMARY:
The purpose of this study is to determine of once identified to the subjects infected with human immunodeficiency virus (positive VIH), to diagnose latent Tuberculosis, and to treat her with isoniazid for six months, measuring the production of Interferon range pre and posttreatment, to evaluate this way the result of the treatment on the immune response

DETAILED DESCRIPTION:
A descriptive analysis of the data will be made. Means and standard deviations for continuous data frequencies for categorical data will be performed. Wilcoxon test Mann-Whitney U test Chi square will be used for frequency analysis of responders Data Analysis and Statistical Software(STATA).

ELIGIBILITY:
Inclusion Criteria:

* Accept to participate. Informed consent.
* Human Immunodeficiency Virus positive test, documented by Western Blot
* Have not received treatment for latent tuberculosis
* Have not been diagnosed pulmonary tuberculosis (Tbp)
* Normal two chest X-rays, Postern-anterior and left lateral.

Exclusion Criteria:

* Active tuberculosis
* Previous diagnosis of tuberculosis
* Antecedent of treatment for active o latent tuberculosis
* Contact with TB patient harboring Multidrug resistance or isoniazid resistant isolates of Mycobacterium tuberculosis.
* Abnormal liver enzyme levels
* Hemoglobin below 8 gr/dl
* Allergy or intolerance to isoniazid
* Peripheral neuropathy
* Ingestion of drugs interacting with isoniazid

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Production of interferon gamma, in response to treatment of latent infection | Before and after treatment intake

CONTACTS AND LOCATIONS:
Overall Officials: José Sifuentes, Doctor, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nitrición Salvador Zubiran (INCMNSZ); Alfredo Ponce-de-León, Doctor, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutrición (INCMNSZ); Maria de Lourdes García-García, Post doctor, Study Director — Instituto Nacional de Salud Publica (INSP); Jose Luis Valdespino-Gómez, MD, Principal Investigator — Laboratorios Nacionales de Biológicos y Reactrivos (BIRMEX); Martha Torres Rojas, Post Doctor, Study Chair — National Institute of Respiratory Diseases (INER)
Locations (2):
- Mexico (2):
  - Instituto Nacional de Salud Publica, México, Cuernavaca Morelos
  - Clínica Especializada CONDESA, Mexico City, D.F